CLINICAL TRIAL: NCT06609876
Title: Thermal Ablation Combined With Low-dose Donafinib for Early Recurrent Hepatocellular Carcinoma: a Multicenter Prospective Study
Brief Title: Donafenib as Adjuvant Therapy Following Ablation for Recurrent HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect1
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; Microwave Ablation; Donafenib; Recurrent Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Transurethral Resection of Prostate; donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal ablation (Experimental): Patients only accepted thermal ablation (microwave ablation,radiofrequency ablation)
  Interventions: Procedure: Thermal ablation
- Microwave ablation plus Donafenib (Experimental): Patients accepted thermal ablation (microwave ablation,radiofrequency ablation) plus Donafenib (100mg, bid)
  Interventions: Procedure: Thermal ablation; Drug: Donafenib

INTERVENTIONS:
Procedure: Thermal ablation — Thermal ablation of tumors
Drug: Donafenib — Donafenib ( 100 mg，bid)
  Arms: Microwave ablation plus Donafenib

SUMMARY:
This study intends to evaluate the efficacy and safety of low-dose adjuvant donafenib after thermal ablation for early recurrent HCC within Milan criteria.

DETAILED DESCRIPTION:
Thermal ablation is available as the major curative treatments for early-stage recurrent HCC. Donafenib was inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma. No study has evaluated low-dose donafenib as adjuvant therapy after thermal ablation. There needs further investigation to explore the efficacy and safety of the combination treatment. Thus, the investigators carried out this prospective, randomized, open-label, phase II trial study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. were aged 18-75 years;
2. had recurrent HCC (RHCC) diagnosed by imaging studies, the first or the second RHCC;
3. RHCC met the Milan criteria, namely single RHCC lesion less than 5 cm in diameter or no more than 3 tumors (each ≤3 cm in diameter);
4. the early RHCC (recurrent time <1 year)
5. patients were unwilling to undergo repeat hepatectomy or liver transplantation;
6. had well-preserved liver function, i.e., Child-Pugh class A or B, and prolonged prothrombin time≤5 s;
7. patients had an Eastern Cooperative Oncology Group performance status score ≤1.
8. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. were under 18 years or over 75 years of age;
2. primary HCC;
3. recurrent HCC beyond Milan criteria;
4. RHCC with metastasis or macrovascular tumor thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Tumor-free survival rate | 24 months
  Progression was defined as progressive disease after thermal ablation by independent radiologic review according to mRECIST or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  OS is the length of time from the date of ablation until death from any cause.
Adverse events | 36 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, Professor, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: No